CLINICAL TRIAL: NCT05050266
Title: Enhancing Mental and Physical Health of Women Through Engagement and Retention (EMPOWER) QUERI 2.0 (QUE 20-028)
Brief Title: Enhancing Mental and Physical Health of Women Veterans
Acronym: EMPOWER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 21-006
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases; Overweight; Obesity; Smoking; Hypertension; Cholesterol; Diabetes Mellitus; Prediabetic State; Pregnancy; Depression, Postpartum; Prevention; Implementation Science; Quality Improvement; Virtual Care
Keywords: Cardiovascular diseases; Overweight; Obesity; Smoking; Hypertension; Cholesterol; Diabetes Mellitus; Prediabetic State; Pregnancy; Depression, Postpartum; Depression; Women; Veterans; Primary Health Care; Mental Health; Patient Participation; Patient Satisfaction; Patient Preference; Physicians, Primary Care; Physicians, Women; Health Behavior; Quality Improvement; Prevention; Heart Disease Risk Factors
MeSH Terms: conditions — Cardiovascular Diseases; Overweight; Obesity; Smoking; Hypertension; Diabetes Mellitus; Prediabetic State; Depression, Postpartum; Depression; Psychological Well-Being; Patient Participation; Patient Satisfaction; Patient Preference; Health Behavior

STUDY DESIGN:
Intervention Model Description: Cluster randomized type 3 hybrid implementation-effectiveness trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- REP (Active Comparator): Replicating Effective Practices (REP) is a lower-intensity implementation strategy with explicit process framework for local tailoring
  Interventions: Behavioral: REP
- EBQI (Experimental): Evidence-Based Quality Improvement (EBQI) is a higher-intensity implementation strategy that entails external facilitation and formal training in quality improvement.
  Interventions: Behavioral: EBQI

INTERVENTIONS:
Behavioral: EBQI — EBQI is a systematic quality improvement method for engaging frontline practices in improvement that introduces "best science" and evidence in the service of operational goals. EBQI has been tested in several VA implementation trials. Sites randomized to EBQI will meet monthly with the implementation support team (i.e., high-intensity).
  Arms: EBQI
Behavioral: REP — The REP framework consists of 4 phases: pre-conditions, pre-implementation, implementation and maintenance/evolution. REP has a strong evidence-base and application in VHA health services research in promoting uptake of EBPs. Sites randomized to REP will meet quarterly with the implementation support team (i.e., low-intensity).
  Arms: REP

SUMMARY:
Women Veterans are the fastest growing segment of VA users. This dramatic growth has created challenges for VA to ensure that appropriate services are available to meet women Veterans' needs, and that they will want and be able to use those services. The EMPOWER QUERI 2.0 Program is a cluster randomized type 3 hybrid implementation-effectiveness trial testing two strategies designed to support implementation and sustainment of evidence-based practices for women Veterans in at least 20 VA facilities from 4 regions.

DETAILED DESCRIPTION:
Women Veterans are the fastest-growing segment of users in the Veterans Health Administration (VA). Their numbers are projected to increase by 73%, from 9.3% to 16.4%, between 2015 and 2043. Despite VA investment in improving care for women Veterans, gender disparities persist in cardiovascular (CV) and diabetes risk factor control. Also, the rate of perinatal depression among women Veterans is higher than that among civilian women, which is of particular concern given the association between perinatal depression and suicidality. Barriers to care for women Veterans include distance to VA care, rurality, competing work and caregiving responsibilities, comorbid mental health issues, and harassment on VA grounds. Improvements are still needed to increase women Veterans' access to and engagement in convenient, safe, evidence-based, patient-centered care that achieves the VA "lane of effort" of Veterans' "lifelong health, well-being, and resilience."

Since its inception in 2015, the Enhancing Mental and Physical health of Women through Engagement and Retention (EMPOWER) QUERI 1.0 team has focused on implementing gender-tailored care models for women Veteran patients. In EMPOWER 1.0 studies, women expressed preferences for gender-specific (women only) care and for virtual care options. Therefore, the EMPOWER 2.0 Impact Goal is to expand access to virtual, evidence-based, preventive lifestyle and mental health services for women Veterans with high-priority health conditions in rural and urban-isolation areas. This cluster randomized type 3 hybrid implementation-effectiveness trial randomized 20 VA sites to one of two implementation strategies, the Replicating Effective Practices (REP) or Evidence-Based Quality Improvement (EBQI), to support implementation and sustainment of evidence-based practices (EBPs). The EBPs focus on preventive lifestyle and mental health care for women Veterans across VA facilities, several of which are rural, low-performing in women's health care, and/or lead sites for high reliability organization. The study team will conduct a mixed methods implementation evaluation to compare the effectiveness of REP and EBQI in terms of: (a) improved access to and rates of engagement in virtual preventive lifestyle and mental health services and improved VA performance metrics for virtual and telehealth care delivery and related clinical outcomes for women Veterans; (b) progression along the Stages of Implementation Completion; (c) adaptation, sense-making, and experiences of EBP implementation among multilevel stakeholders; and (d) cost and return on investment.

On 8/15/23, as part of our 12 month registration update corrected the primary outcomes to accurately reflect the randomized trial and analyses design. The cluster randomized trial will evaluate the effectiveness of two implementation strategies (REP and EBQI) in implementing evidence-based practices (EBPs) for preventive services. Although we are implementing three evidence-based practices (DPP, TLC and ROSE), the EBPs are combined for each of the trial's two primary outcomes (access and engagement).

ELIGIBILITY:
Inclusion Criteria:

This study is recruiting VA sites - not individual patients. Prior to randomization, the study team will work with sites to ensure they have met the preconditions necessary to enroll in the study, which includes VISN, regional and/or facility level leadership support for participation.

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Access to virtual care for preventive services | 12 months
  Proportion of eligible women Veterans who enroll in virtual DPP, TLC, or ROSE at each site
Engagement in virtual care for preventive services | 12 months
  Proportion of eligible women Veterans who attend 1 or more virtual DPP, TLC, or ROSE sessions at each site

SECONDARY OUTCOMES:
Participation and engagement: DPP | 6 and 12 months
  average # of sessions attended by women Veterans who enrolled in DPP at each site
Participation and engagement: DPP | 6 and 12 months
  proportion who completed >9 and >16 sessions among women Veterans who enrolled in DPP at each site
Participation and engagement: DPP | 6 and 12 months
  % weight change among women Veterans who enrolled in DPP at each site
Participation and engagement: TLC | 6 months
  average # of TLC sessions completed among women Veterans who enrolled in TLC at each site
Participation and engagement: TLC | 6 months
  % with health behavioral goal among women Veterans who enrolled in TLC at each site
Participation and engagement: TLC | 6 months
  % with behavioral change (physical activity, diet: fruit, vegetable and sugary beverage intake, stress and coping, and weight) at each site
Participation and engagement: ROSE | 6 months
  average # of ROSE sessions completed at each site

CONTACTS AND LOCATIONS:
Overall Officials: Alison B Hamilton, PhD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Data sets underlying all publications resulting from the proposed research will not be shared outside VA, except as required under the Freedom of Information Act (FOIA), because VHA policy would prohibit re-disclosure.

REFERENCES:
- [Derived] Finley EP, Hamilton AB, Canelo I, Jackson SS, Lesser R, Oberman RS, Yosef J, Chrystal JG, Fletcher EH, Bean-Mayberry B, Moin T, Farmer MM, Lang AJ. Collaborative tailoring of the Reach Out, Stay Strong Essentials (ROSE) program for pregnant veterans in the U.S. Veterans Health Administration: a qualitative case study of contextual conditions and adaptations. BMC Health Serv Res. 2025 May 23;25(1):746. doi: 10.1186/s12913-025-12871-x. PMID 40410822
- [Derived] Malone A, Clair K, Chanfreau C, Bean-Mayberry B, Oberman R, Lesser R, Knight C, Finley E, Hamilton A, Farmer MM, Moin T. Predictors of enrollment in a virtual diabetes prevention program among women veterans: a retrospective analysis. BMC Womens Health. 2024 Aug 24;24(1):465. doi: 10.1186/s12905-024-03314-6. PMID 39180036
- [Derived] Finley EP, Chrystal JG, Gable AR, Fletcher EH, Palma A, Canelo I, Oberman RS, Jackson SS, Lesser R, Moin T, Bean-Mayberry B, Farmer MM, Hamilton A. The Rapid Implementation Feedback (RIF) report: real-time synthesis of qualitative data for proactive implementation planning and tailoring. Implement Sci Commun. 2024 Jun 21;5(1):69. doi: 10.1186/s43058-024-00605-9. PMID 38907331
- [Derived] Hamilton AB, Finley EP, Bean-Mayberry B, Lang A, Haskell SG, Moin T, Farmer MM; EMPOWER QUERI Team. Enhancing Mental and Physical Health of Women through Engagement and Retention (EMPOWER) 2.0 QUERI: study protocol for a cluster-randomized hybrid type 3 effectiveness-implementation trial. Implement Sci Commun. 2023 Mar 8;4(1):23. doi: 10.1186/s43058-022-00389-w. PMID 36890587
- See also: project executive summary — https://www.queri.research.va.gov/centers/EMPOWER.pdf